CLINICAL TRIAL: NCT04780802
Title: Balloon Assisted Transarterial Therapy for Hepatocellular Carcinoma: a Study on the Proof of Treatment Concept and Exploration of Selection Criteria for Clinical Application
Brief Title: Balloon Assisted Transarterial Therapy for Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-20-13
Record Dates: First submitted 2020-11-30; First posted 2021-03-04 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ballloon catheter (Other): Balloon-assisted transarterial therapy will be performed in the first treatment session only
  Interventions: Procedure: The balloon catheter is placed at the various arterial feeders of the tumor

INTERVENTIONS:
Procedure: The balloon catheter is placed at the various arterial feeders of the tumor — use of a balloon catheter for providing balloon occlusion, in addition to the standard microcatheter for drug delivery, both catheters are to be placed in parallel through a single guide catheter. Only one arterial puncture wound is involved. The inflated balloon provides temporary occlusion of all arterial tumor feeders except for the one which is selectively catheterized with a microcatheter for delivery of the therapeutic agent. The therapeutic agent consists of Lipiodol mixed with a chemotherapeutic drug, it is delivered through the microcatheter under fluoroscopic control.

SUMMARY:
To prove the treatment concept of the use of balloon assistance in transarterial therapy for HCC.

DETAILED DESCRIPTION:
Transcatheter arterial chemoembolization (TACE) has been playing an important role in the treatment algorithm for patients with multifocal or large intrahepatic lesions of hepatocellular carcinoma (HCC) not eligible for surgical resection, transplantation, or local ablative therapy. The use of balloon assisted TACE has been proposed recently and it could be one of the possible ways to improve the effectiveness of drug delivery to the target tumor and therefore leading to improved treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age above 18 years
2. Patients who are indicated for transarterial treatment for HCC
3. Child-Pugh A or B cirrhosis
4. Eastern Cooperative Oncology Group performance score 0 or 1
5. BCLC A or B
6. No previous treatment with liver resection, ablation, chemotherapy, radiotherapy or transarterial embolization (with or without chemotherapy),
7. HCC diagnosed by typical enhancement patterns on cross sectional imaging or histology.
8. No extra-hepatic involvement on non-enhanced CT thorax and triphasic contrast enhanced CT abdomen.
9. No invasion of portal vein or hepatic vein
10. Massive expansive tumor morphology with measurable lesion on CT (characterized by well-defined spherical or globular configuration, with or without tumor capsule or satellite lesions)
11. Total tumor mass < 50% liver volume
12. Size of any individual tumor <= 7cm in largest dimension
13. Serum creatinine < 130 umol/L or Creatinine clearance > 55 ml/min.

Exclusion Criteria:

1. Concurrent ischemic heart disease or heart failure
2. History of asthma, chronic obstructive airway disease or respiratory decompensation.
3. History of acute tumor rupture presenting with hemo-peritoneum
4. Biliary obstruction not amenable to percutaneous or endoscopic drainage
5. Child-Pugh C cirrhosis
6. History of hepatic encephalopathy
7. Intractable ascites not controllable by medical therapy
8. History of variceal bleeding within last 3 months
9. Serum total bilirubin level > 50 umol/L
10. Serum albumin level < 26 g/L
11. INR > 1.3
12. Infiltrative tumor morphology (characterized by ill- defined tumor margin and amorphous configuration) or diffuse tumor morphology (characterized by large number of small nodules)
13. Arterio-portal venous shunt affecting >1 hepatic segment on CT
14. Arterial-hepatic venous shunt with hepatic vein opacified in arterial phase on CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The change in hemodynamics of arterial blood supply to HCC tumors | immediately after completion of procedure
  The change in number of feeding arteries
The change in the perfusion pattern of HCC tumors | immediately after completion of procedure
  The change in perfusion pressure.

SECONDARY OUTCOMES:
Tumor response | 3 months
  Tumor response by CT such as complete response according to European Association for the Study of the Liver (EASL) necrosis guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Professor, Principal Investigator — DIIR, CUHK, Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No